CLINICAL TRIAL: NCT03442868
Title: Efficacy of Non-Invasive Brain Stimulation on Dual-Task Walking After Stroke: A Repetitive Transcranial Magnetic Stimulation (rTMS) Study
Brief Title: Non-invasive Brain Stimulation (NIBS) and Dual-task Walking After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Hui Ting Goh, Assistant Professor, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19219
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- High frequency rTMS (Experimental): High frequency rTMS will be applied to different neural loci based on the randomized sessions.
  Interventions: Device: high frequency rTMS

INTERVENTIONS:
Device: high frequency rTMS — Participants receive 16 minutes (5Hz, 24 10-second trains with a inter-train interval of 30s) of high frequency rTMS applied to either primary motor cortex (M1), supplementary motor area (SMA) and dorsolateral prefrontal cortex (DLPFC) at different sessions. Walking performance is evaluated before and after the brain stimulation.

SUMMARY:
The study aims to identify neural locus critical for dual-task walking (walking and talking) in individuals with stroke. To achieve this aim, the investigators apply repetitive transcranial magnetic stimulation (rTMS) to different parts of the brain and evaluate the effects of brain stimulation on dual-task walking speed.

DETAILED DESCRIPTION:
This study will enroll 12 individuals with a stroke at least 6 months ago. Participants will be tested across 3 sessions and each session will be approximately 1 week apart from each other. During testing, participants will be asked to walk under two conditions: single- and dual-task conditions. Under the single-task condition, participants walk on a instrumented mat such that their gait performance will be captured. Under the dual-task condition, participants walk on the mat while performing a counting backward task. The walking assessment is followed by a 12 minute non-invasive brain stimulation using high frequency rTMS. Another walking assessment will be conducted right after the brain stimulation session. High frequency rTMS will be applied to different neural loci, namely primary motor cortex (M1), supplementary motor area (SMA), and dorsolateral prefrontal cortex (DLPFC). The walking speed under two different conditions will be compared before and after brain stimulation to different neural loci.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Diagnosis of Left hemispheric stroke at least 6 months ago
3. First time stroke OR complete gait recovery from prior stroke
4. Able to walk independently for at least 10 meters with or without walking aids
5. Have at least minimal movements (> 5 degree of motion) at the affected ankle
6. Score > 26 on Mini Mental State Exam (MMSE)
7. Ability to participate in the informed consent process

Exclusion Criteria:

1. Diagnosis of other neurological conditions, such as Parkinson Disease, Alzheimer, Spinal Cord Injury, Multiple Sclerosis
2. Other comorbidities which could interfere with gait (i.e. amputation, severe osteoarthritis)
3. Unstable clinical conditions
4. Non-ambulatory prior to onset of stroke
5. History of significant head trauma
6. Electrical, magnetic, or mechanical implantation: cardiac pacemakers or intracerebral vascular clip
7. Metal implantation in the oral cavity, head/neck area and lower extremity
8. Pregnancy
9. History of seizures or unexplained loss of consciousness
10. Immediate family member with epilepsy
11. Use of seizure threshold lowering medicine
12. Current abuse of alcohol or drugs
13. Anticipated inability to complete the study
14. History of psychiatric illness requiring medication control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ting Goh, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Dallas Fort Worth metro area. Recruitment started in October 2016 and last participant was enrolled in Oct 2018.
Groups:
- High Frequency Repetitive Transcranial Magnetic Stimulation (rTMS): High frequency rTMS will be applied to different neural loci based on the randomized sessions.
  high frequency rTMS: Participants receive 16 minutes (5Hz, 24 10-second trains with a inter-train interval of 30s) of high frequency rTMS applied to either primary motor cortex, supplementary motor areas and dorsolateral prefrontal cortex at different sessions. Walking performance is evaluated before and after the brain stimulation.
Period: Overall Study
Arm/Group | High Frequency Repetitive Transcranial Magnetic Stimulation (rTMS)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- High Frequency rTMS: High frequency rTMS will be applied to different neural loci based on the randomized sessions.
  high frequency rTMS: Participants receive 16 minutes (5Hz, 24 10-second trains with a inter-train interval of 30s) of high frequency rTMS applied to either primary motor cortex, supplementary motor areas and dorsolateral prefrontal cortex at different sessions. Walking performance is evaluated before and after the brain stimulation.
Arm/Group | High Frequency rTMS
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Gait Speed
Description: gait speed in m/s will be captured using GaitRite gait assessment walkway
Time Frame: before and 10 minutes after the non-invasive brain stimulation
Population: Changes in gait speed under the dual-task conditions were compared across the 3 visits.
Measure: Mean (Standard Error); unit: m/s
Arm/Group | High Frequency rTMS
Number analyzed (Participants) | 15
m/s
  Primary motor cortex (M1) | -0.49 (1.66)
  Supplementary motor area (SMA) | -0.80 (2.64)
  Dorsolateral prefrontal cortex (DLPFC) | 5.49 (2.19)

2. Secondary Outcome: Change in Step Lengths
Description: Step lengths in centimeter (cm) will be captured using GaitRite gait assessment walkway
Time Frame: before and 10 minutes after the non-invasive brain stimulation
Population: Changes in right (R) and left (L) step lengths after repetitive transcranial magnetic stimulation (rTMS) applied to dorsolateral prefrontal cortex (DLPFC)
Measure: Mean (Standard Error); unit: centimeter (cm)
Arm/Group | High Frequency rTMS
Number analyzed (Participants) | 15
centimeter (cm)
  Changes in R step length after rTMS to DLPFC | 2.24 (1.02)
  Changes in L step length after rTMS to DLPFC | 1.38 (1.13)

3. Secondary Outcome: Change in Single Support Times
Description: Single support times (in % of gait cycle) will be captured using GaitRite gait assessment walkway
Time Frame: before and 10 minutes after the non-invasive brain stimulation
Population: Changes in right (R) and left (L) single support time after repetitive transcranial magnetic stimulation (rTMS) applied to dorsolateral prefrontal cortex (DLPFC)
Measure: Mean (Standard Error); unit: percentage of gait cycle
Arm/Group | High Frequency rTMS
Number analyzed (Participants) | 15
percentage of gait cycle
  changes in R single support after rTMS to DLPFC | 0.63 (1.87)
  changes in L single support after rTMS | 2.50 (1.11)

4. Secondary Outcome: Change in Counting Task Performance
Description: number of correct responses in counting backward task
Time Frame: before and 10 minutes after the non-invasive brain stimulation
Population: number of correct response under the dual-task conditions before and after the rTMS
Measure: Mean (Standard Error); unit: number of correct responses
Arm/Group | High Frequency rTMS
Number analyzed (Participants) | 15
number of correct responses
  Primary motor cortex (M1) | -0.18 (0.83)
  Supplementary motor area (SMA) | -0.59 (0.66)
  Dorsolateral prefrontal cortex (DLPFC) | -0.65 (0.74)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | High Frequency rTMS
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Frequency rTMS (N=15)
Headache (General disorders) | 1 (1) — 1 participant reported mild headache after stimulation. The headache was resolved about 2 hours after the session ended.
Infection (Infections and infestations) | 1 (1) — 1 participant was admitted to the hospital between the1st and the 2nd visit due to a lung infection. The event was deemed unrelated to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT03442868/Prot_SAP_000.pdf